CLINICAL TRIAL: NCT05017896
Title: Prediction of Acute Kidney Injury After Operation of Acute Type A Aortic Dissection Based on Multimodal Model
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020SDUCRCC031
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Aneurysm, Dissecting; Acute Kidney Injury
MeSH Terms: conditions — Aortic Dissection; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Perfusion
  Interventions: Diagnostic Test: Normal CT Renal Perfusion imaging indexes
- Low Perfusion
  Interventions: Diagnostic Test: Low CT Renal Perfusion imaging indexes

INTERVENTIONS:
Diagnostic Test: Normal CT Renal Perfusion imaging indexes — A CT imaging which indicates the status of renal perfusion is normal.
  Groups: Normal Perfusion
Diagnostic Test: Low CT Renal Perfusion imaging indexes — A CT imaging which indicates the status of renal perfusion is low.
  Groups: Low Perfusion

SUMMARY:
Acute kidney injury is one of the most common postoperative complications of acute type A aortic dissection, which is closely related to early postoperative death. Early prevention, early diagnosis and early treatment are the key to improve the prognosis of such patients. It has been a hot topic in clinical research for a long time. Previous reports revealed a series of risk factors for acute kidney injury after aortic dissection, but limited by research design and single modal data, high quality studies were rare. The purpose of this study is to further clarify the risk factors by studying the relationship between preoperative CT renal perfusion imaging indexes and postoperative acute kidney injury; establish and externally verify the multimodal radiomics prediction model for acute kidney injury after operation of aortic dissection combining with preoperative CT renal perfusion imaging and CT angiography information by analysis methods of information fusion, feature engineering and radiomics, so as to guide the follow-up clinical practice, improve the prognosis of such patients and save medical resources.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old
2. Acute type A aortic dissection diagnosed by CT angiography
3. Sign informed consent

Exclusion Criteria:

1. History of chronic kidney disease
2. History of cardiovascular operation
3. Acute kidney injury has occurred before operation
4. Pregnancy status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients sufferred acute type A aortic dissection.
Sampling Method: Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury after operation | From date of operation until the date of acute kidney injury or date of death from any cause, whichever came first, assessed up to 30 days.
  Yes; No

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zhao, Principal Investigator — Department of cardiac surgery, Qilu Hospital, Shandong University

IPD SHARING:
Plan to Share IPD: Undecided